CLINICAL TRIAL: NCT04852107
Title: Prospective, Randomized, Double Blinded Crossover Study Comparing Spinal Cord Stimulation (SCS) vs Dorsal Root Ganglion Stimulation (DRGS) vs Association of Both (DUAL) in Patients With Refractory Chronic Lower Limb Neuropathic Pain and/or Back Neuropathic Pain
Brief Title: Comparative Study in Patients With Refractory Chronic Lower Limb Neuropathic Pain and/or Back Neuropathic Pain.
Acronym: BOOST DRG
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Sponsor decision
Sponsor: Poitiers University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Screening
Other Study IDs: 2020-A03020-39
Record Dates: First submitted 2021-03-26; First posted 2021-04-21 (Actual); Last update posted 2023-01-13 (Actual); Status verified 2023-01

CONDITIONS: Pain, Neuropathic
Keywords: Dorsal Root Ganglion; Spinal Cord Stimulation
MeSH Terms: conditions — Neuralgia | interventions — Spinal Cord Stimulation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- SCS/ DRGS/DUAL /Dual* (Active Comparator)
  Interventions: Other: Spinal Cord Stimulation, association of both (DUAL), Dorsal Root Ganglion stimulation
- SCS/DUAL/DRGS/DRGS* (Active Comparator)
  Interventions: Other: Spinal Cord Stimulation, association of both (DUAL), Dorsal Root Ganglion stimulation
- DRGS/SCS/DUAL/DUAL* (Active Comparator)
  Interventions: Other: Spinal Cord Stimulation, association of both (DUAL), Dorsal Root Ganglion stimulation
- DRGS/DUAL/SCS/SCS* (Active Comparator)
  Interventions: Other: Spinal Cord Stimulation, association of both (DUAL), Dorsal Root Ganglion stimulation
- Dual/DRGS/SCS/SCS* (Active Comparator)
  Interventions: Other: Spinal Cord Stimulation, association of both (DUAL), Dorsal Root Ganglion stimulation
- Dual/SCS/DRGS/DRGS* (Active Comparator)
  Interventions: Other: Spinal Cord Stimulation, association of both (DUAL), Dorsal Root Ganglion stimulation

INTERVENTIONS:
Other: Spinal Cord Stimulation, association of both (DUAL), Dorsal Root Ganglion stimulation — Lead Implantation which will be conducted in 2 steps:
  1. Lead implantation: 8-contact SCS percutaneous lead on SC and 8-contact lead on DRG.
  2. Neurostimulation trial phase (Mode DUAL). IPG implantation + Randomization + 1st leads programming (SC, DRG or DUAL stimulation according to randomization sequence).
  2nd leads programming (SC, DRG or DUAL stimulation according to randomization sequence). 3rd leads programming (SC, DRG or DUAL stimulation according to randomization sequence). All patients will be switched to Burst waveform for a 1- month follow-up period while keeping the last allocated stimulation type in the randomized crossover arm.

SUMMARY:
Neuropathic pain is described as a "pain initiated or caused by a primary lesion or dysfunction in the nervous system". It is thus often a chronic affection, as a difficult-to-treat condition. As such, there is growing proportion of patients with inefficient pain relief. The prevalence of chronic neuropathic pain has been estimated from 6.9 to 10% in the general population and represents a heavy financial burden for the health care systems. Spinal Cord Stimulation (SCS) is a well-established therapy to alleviate severe intractable neuropathic pain (SCS is a reversible treatment option which leads to improve pain relief and quality of life Using conventional SCS, the prerequisite to target any pain relief is to obtain an appropriate coverage of the painful area with induced paresthesia.

Despite its effectiveness, conventional SCS has some limitations (Selectivity, Energy consumption …) and in order to address these limitations and challenges, medical devices and neuromodulation industries have developed the Dorsal Root Ganglion (DRG) stimulation. DRG stimulation appears to be a promising technology that can be proposed to patients with chronic neuropathic pain for several reasons: DRG stimulation has shown promising results in pathologies generating focal pain with more selectively than SCS, lead localization appeared to be less discriminative than SCS. Consequently, DRG seems more stable and efficient to relief pain with lower energy consumption than SCS (therapy can be delivered with very low amplitude compared to SCS).

Last but not least, Abbott technology has moved forward to Burst stimulation a couple of years ago and validated this new way of delivering electrical stimulation through several major publications. To our knowledge, applying new waveforms to DRG has not been yet validated. This will represent a fantastic opportunity to refine the design of the next generation of Internal Pulse Generators (IPGs).

To date, the baseline study comparing DRG stimulation to SCS is the ACCURATE study. This is a high quality prospective, multicenter, randomized comparative trial conducted in 152 patients implanted with either SCS or DRG stimulation system. Although ACCURATE study is well designed, it has some limitations.

To bridge this gap, the investigators propose to conduct a randomized controlled trial (RCT) with a crossover design, where SCS and DRG stimulation will be used within patient in three conditions: (i) SCS alone, (ii) DRG stimulation alone (DRGS), (iii) combination of SCS and DRGS (DUAL).

Our goal will be to compare SCS vs DRGS vs DUAL therapies in order to establish the superiority of DRG stimulation over SCS in a crossover design, assess the added value of hybrid stimulation (DUAL) over the separate standalone stimulation types, compare the different cortical pathways involved in both techniques, by functional imaging, incl. MRI, analyze energy consumption by optimizing neural targeting. assess the added value of applying Burst on these different targets, after a 3-month follow-up and to reinforce the perception of neurostimulation techniques through the pain community, as the investigators will demonstrate their benefits on pain relief, functional capacity and quality of life, with objectives measures and a randomized design. This study represents a unique opportunity to boost the rationale of SCS/DRGS since each arm of treatment will be blinded for the patient and the implanter.

ELIGIBILITY:
Inclusion Criteria:

* Subject has ≥ 18 years and ≤ 80 years
* Subject has a VAS ≥ 5
* Subject has refractory chronic lower limbs neuropathic pain (e.g. diabetic foot peripheral neuropathy, foot peripheral neuropathy, ankle peripheral neuropathy) or/and neuropathic back pain for at least 6 months
* Subject has stable pain for at least 30 days
* Pain medication(s) dosage(s) is/are stable for at least 30 days
* Subject is refractory to other treatment modalities (e.g. Medication, psychological therapies, pain interventions, surgery)
* Subject is eligible for SCS after a pre-implantation assessment by a multidisciplinary team, as described by the French National Authority for Health
* Subject understands and accepts constraints of the study.
* Patient covered by French national health insurance.
* Subject has given written consent to the study after having received clear and complete information

Non inclusion criteria:

* Subject has a coagulation disorder
* Subject is or has been treated with SCS, subcutaneous or peripheral nerve stimulation, an intrathecal drug delivery system
* Subject has had corticosteroid therapy within the past 30 days
* Subject has had radiofrequency therapy within the past 3 months
* Subject has been diagnosed with cancer in the past 2 years
* Subject has had a spinal surgery within the past 6 months
* Subjects requiring closer protection, i.e. minors, pregnant women, nursing mothers, subjects deprived of their freedom by a court or administrative decision, subjects admitted to a health or social welfare establishment, major subjects under legal protection, and finally patients in an emergency setting
* Simultaneous participation to any interventional study on health product or any study able to interfere with the current study endpoints.
* Pregnant or breastfeeding women, women at age to procreate and not using effective contraception
* Brain MRI contraindication

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2021-08-20 (Actual); Primary Completion 2022-12-15 (Actual); Study Completion 2022-12-15 (Actual)

PRIMARY OUTCOMES:
To compare pain relief with SCS vs DRGS vs association of both (DUAL) in patients with chronic lower limb neuropathic pain and/or back neuropathic pain following each stimulation modality within a 3-month crossover period. | 3 Months
  Proportion of patients having a reduction of 50% on the Visual Analogic Scale (VAS) score (0-No pain/10-worst pain imaginable) (assessed with a 5-day pain diary) between baseline (before leads implantation) and after the end of each period of crossover phase.

SECONDARY OUTCOMES:
Mean pain intensity score | 12 months
  Pain intensity will be assessed using the Visual Analogic Scale (VAS) score (0-No pain/10-worst pain imaginable) at Lead Implantation Visit, M0, M1, M2, M3, M4, M6 and M12.
Mean pain surface (cm²) | 12 months
  Global Pain surface (cm²) measured using a pain mapping tool at Lead Implantation Visit, M0, M1, M2, M3, M4, M6 and M12.

OTHER OUTCOMES:
Mean pain surface for each pain intensity (cm²) | 12 months
  Pain intensities associated with the surface measurements measured using a pain mapping tool at Lead Implantation Visit, M0, M1, M2, M3, M4, M6 and M12.
Mean lead performance | 12 months
  Lead performance is measured as the percentage of pain covered with paresthesia at Lead Implantation Visit, M0, M1, M2, M3, M4, M6 and M12.
Mean lead selectivity | 12 months
  Lead selectivity is measured as the percentage of paresthesia covering pain at Lead Implantation Visit, M0, M1, M2, M3, M4, M6 and M12.
Mean discomfort associated with paresthesia. | 12 months
  Discomfort will be assessed using a 11-points NRS (0-no discomfort/10-severe discomfort) at sitting, standing and lying down at M1, M2, M3, M4, M6 and M12.
Mean health-related quality of life score | 12 months
  Health-related quality of life will be assessed using the EuroQol 5-Dimensions index (0-worst imaginable health condition/1-Best Health condition) at Inclusion Visit, M0, M1, M2, M3, M4, M6 and M12.
Mean functional disability score | 12 months
  Functional disability will be assessed using Oswestry Disability Index percentage (0%-the patient can cope with most living activities/100%- These patients are either bed-bound or exaggerating their symptoms.) at Inclusion Visit, M0, M1, M2, M3, M4, M6 and M12.
Mean anxiety and depression scores | 12 months
  Anxiety and depression will be assessed using the Hospital Anxiety and Depression Scale scores (0 to 14 : no anxiety or depressive disorders/ 15 to 42: existence of anxiety-depressive disorders.) at Inclusion Visit, M0, M1, M2, M3, M4, M6 and M12.
Mean catastrophizing score | 12 months
  Catastrophizing will be assessed using Pain Catastrophizing Scale scores (0 to 52) at Inclusion Visit, M0, M1, M2, M3, M4, M6 and M12.
Patient satisfaction | 12 months
  Satisfaction will be assessed using the Patient Global Impression of Change scale scores (0-No change or it gets worse/ 6-Significantly better, a considerable improvement that makes all the difference) at M0, M1, M2, M3, M4, M6 and M12.
Percentage of responders as defined by the following composite stimulation efficacy score | 12 months
  Stimulation efficacy is defined as having at least three of the criteria listed below, 12 months following IPG implantation (patients with a negative lead trial will be considered as nonresponders).
  * Regaining functional capacity: Having at least a 30% decrease in the ODI score.
  * Adequate global pain relief: Having at least a 50% decrease in the VAS.
  * Improvement in quality of life: Having at least a 0.2 points increase in the EQ-5D index.
  * Decrease in psychological distress: Having a decrease of 1.4 points in the HADS depression score.
  * 30% decrease in pain surface (percentage of cm²)
  * Having a PGIC score of at least 6.
  * Drug intake: drug intake will be measured using the Medication Quantification Scale III (MQS) and a reduction of 3.4 points will be considered as meaningful.
Rate of adverse events | 12 months
  Safety will be evaluated by the rate of Adverse Events (AE), Serious Adverse Events (SAE) and device deficiencies from Inclusion to M12.
EEG characteristics will be collected, ratio between the dorsal anterior cingulate cortex and pregenual anterior cingulate cortex/ventromedial prefrontal cortex will be measured. | 4 months
  Ratio between the dorsal anterior cingulate cortex (dACC) and pregenual anterior cingulate cortex/ventromedial prefrontal cortex (pgACC/vmPFC) will be measured at inclusion, M3 and M4.
fMRI characteristics will be collected using Blood Oxygen Level Dependent (BOLD) functional Magnetic Resonance Imaging (fMRI). | 4 months
  Stimulations effects on brain activity will be studied using Blood Oxygen Level Dependent (BOLD) functional Magnetic Resonance Imaging (fMRI). BOLD fMRI response in pain related brain regions such as primary/secondary somatosensory cortex, retrosplenial granular cortex, thalamus, caudate putamen, nucleus accumbens, globus pallidus, and amygdala will be assessed at inclusion, M3 and M4.

CONTACTS AND LOCATIONS:
Overall Officials: Philippe RIGOARD, MD, PhD, Principal Investigator — Poitiers Hospital University
Locations (1):
- Poitiers University Hospital, Poitiers, France